CLINICAL TRIAL: NCT05246085
Title: Evaluating Adrenal Insufficiency in Adults With Eosinophilic Esophagitis on Chronic Swallowed Topical Steroids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: Protocol 21-4826; UL1TR001082 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-02-18 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steroid: Subjects who take chronic swallowed topical steroids (i.e. budesonide or fluticasone) will be enrolled in the steroid cohort.
  Interventions: Diagnostic Test: Cortisol level
- Proton pump inhibitor: Subjects who take chronic proton pump inhibitors will be enrolled in the proton pump inhibitor cohort.
  Interventions: Diagnostic Test: Cortisol level

INTERVENTIONS:
Diagnostic Test: Cortisol level — Cortisol levels will be checked in both groups to screen for adrenal insufficiency.

SUMMARY:
Eosinophilic esophagitis (EoE), a chronic inflammatory disease of the esophagus, is a clinical and financial burden to patients if left untreated. Often the natural history of the disease includes development of fibrosis and stricturing of the esophagus, acute food impactions, unplanned emergency room visits, and invasive procedures such as endoscopy. Currently there are no Food and Drug Administration (FDA) approved medications for the treatment of EoE. As such, pharmacologic options approved for use in asthma are used for treatment of EoE and include proton pump inhibitors and swallowed topical steroids. These medications are prescribed chronically as EoE is considered a lifelong disease. Chronic administration of exogenous steroids, when given in inhaled or systemic preparations, can lead to adrenal insufficiency (AI). AI is seen in 7.8% of patients receiving chronic inhaled steroids and 48.7% of patients receiving chronic systemic steroids. The administration of steroids in EoE is unique, as patients typically swallow topical preparations of the drug. The risk of secondary AI from taking swallowed topical steroids is currently unknown, as there has been no study in an adult population assessing this risk as a primary endpoint. Pediatric studies of patients with EoE have shown the risk of AI from swallowed topical steroids to be 5-10%. Based on the risk of AI with inhaled steroids (7.8% prevalence) and the prevalence of AI from swallowed topical steroids in pediatric populations (5-10%), we hypothesize that the risk with swallowed topical steroids is >5%. This could warrant consideration of screening given the potentially serious consequences of undiagnosed AI. To address this hypothesis, this project aims to define the prevalence of developing AI in adults with EoE taking swallowed topical steroids and compare that prevalence to a similar control population of adults with EoE who are taking proton pump inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* 300 adult male or female patients between 18 and 85 years of age with a diagnosis of eosinophilic esophagitis who have been on swallowed topical steroids or proton pump inhibitor therapy (any dosing) for at least 3 months.

Exclusion Criteria:

* We will exclude control patients on proton pump inhibitor therapy if they have used any form of exogenous steroids within the past one year.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled during visits at the University of Colorado Anschutz Medical Campus gastroenterology clinic and endoscopy center.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of adrenal insufficiency | 1 year
  Low cortisol level that is confirmed using an adrenocorticotropic hormone stimulation test.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli DeLay, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT05246085/Prot_SAP_000.pdf